CLINICAL TRIAL: NCT03796117
Title: Neuromuscular Parameters, Current Intensity and Discomfort Level Between Pulsed Current and Russian Current in Healthy Young Subjects.
Brief Title: Pulsed Current Versus Russian Current Effects in Healthy Young Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 3.064.351
Record Dates: First submitted 2018-12-24; First posted 2019-01-08 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Healthy Young; Electric Stimulation Therapy
Keywords: Muscle Strength; Fatigue; Neuromuscular efficiency; Discomfort level; Electric Stimulation
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1: healthy young (Experimental): Participants receive two interventions (Pulsed Current - PC, or Russian Current - RC) in a specific order, according to randomization. Evoked torque, discomfort level, current intensity, neuromuscular efficiency, clinical efficiency and fatigability level will be evaluated.
  Interventions: Device: Pulsed current; Device: Russian Current
- Experimental Group 2: healthy young (Experimental): Participants receive two interventions (Pulsed Current - PC, or Russian Current - RC) in a specific order, according to randomization. Evoked torque, discomfort level, current intensity, neuromuscular efficiency, clinical efficiency and fatigability level will be evaluated.
  Interventions: Device: Pulsed current; Device: Russian Current

INTERVENTIONS:
Device: Pulsed current — For stage 1 of the study, which corresponds to analysis of the evoked torque, evaluation of the discomfort level, current intensity, analysis of neuromuscular efficiency and clinical efficiency, 2 configurations (PC1 and PC2) will be used.
  PC1, will be set at a frequency of 100 Hz, phase duration of 1000 microseconds, ON-OFF time of 5s:10s.
  PC2, will be set at a frequency of 100 Hz, phase duration of 200 microseconds ON-OFF time of 5s:10s.
  For stage 2 of the study, which corresponds to the analysis of the fatigability level, only the PC1 configuration will be used.
Device: Russian Current — For stage 1 of the study, which corresponds to analysis of the evoked torque, discomfort level, current intensity, neuromuscular efficiency and clinical efficiency, 2 configurations (RC1 and RC2) will be used.
  RC1, will be set to a frequency of 100 Hz, burst duty cycle of 20%, ON-OFF time of 5s:10s.
  RC2, will be set at a frequency of 100 Hz, burst duty cycle of 50%, ON-OFF time of 5s:10s.
  For stage 2 of the study, which corresponds to the analysis of the fatigability level, only the RC2 configuration will be used.

SUMMARY:
Low frequency pulsed current (PC) and medium frequency alternating current (Russian current - RC, 2.5 kHz) have been largely studied due to their clinical use. However, it is not clear which current is the most efficient due to the existente literature conflicts.Therefore, the purpose of this study is to compare the neuromuscular efficiency, evoked torque, current intensity, fatigability and level of discomfort between the PC and the RC in healthy young. The current types will be tested in the same participant by the intervention sequences randomization. On the first, second, third and fourth days, the maximum voluntary isometric contraction (MVIC), the current intensity level, discomfort level, evoked torque, and clinical and neuromuscular efficiency of each current will be evaluated. Anthropometric measurements will also be assessed on the first day. In addition, the current intensity required to produce a torque level of 20% of the MVIC, the current intensity required to generate a torque of 40 Nm and the maximum intensity tolerated by the participant will be evaluated. Three contractions will be recorded in each condition, and the level of discomfort will be assessed during the evoked contractions. Evoked torque will be evaluated at the maximum tolerated intensity level using the isokinetic dynamometer. Clinical and neuromuscular efficiency will be evaluated (1) at the current intensity necessary to evoke 20% MVIC, (2) at the current intensity necessary to generate 40 Nm, and (3) at the maximum tolerated current intensity. On the fifth and sixth days, muscle fatigue induced by the diferente current types will be evaluated. Fatigue will be evaluated with sufficient current intensity to generate 20% of the MVIC. MVIC will be performed before and after the fatigue protocol, and the fatigue will be determined by the relative variation of the MVIC before and after the fatigue protocol. Fatigue will also be evaluated through the evoked torque variation between the first and the last minute of the fatigue protocol, as well as by the total work generated in each protocol. Neuromuscular efficiency will be evaluated before and immediately after the protocol through (1) the ratio between input NMES current intensity and output evoked torque, (2) total work (area under the evoked force by time curves) generated during the fatigue protocol, and (3) by the changes in muscle architecture from rest to evoked contraction at the maximal current intensity.

DETAILED DESCRIPTION:
This study is characterized by a quantitative approach, with a randomized crossover clinical study design, blinded to evaluators and participants. The objective is to compare the neuromuscular and clinical efficiency, evoked torque, current intensity, fatigue and discomfort level between the low frequency biphasic pulsed current (PC) and the median frequency sinusoidal alternating Russian current (RC) in healthy young participants. The effect of the two neuromuscular electrical stimulation (NMES) current types on the cited variables will be evaluated in the same participant, by means of the randomization of the interventions sequences for each participant. The evaluation protocols will be performed by 2 blinded raters for the current type and for the outcome variables. A blinded evaluator to the study will randomize the current type, which will be applied on the different evaluation days, through a lottery using opaque envelopes. A researcher blinded to the study groups will analyze the data. Participants will be blinded to the current type will be receiving. The evaluations will be performed in six days, and a minimum interval of 7 days will be observed between the evaluation days. On the first, second, third and fourth days, characterized as Stage 1, the currents' intensity levels, discomfort level, evoked torque, and neuromuscular and clinical efficiency of each randomized current will be evaluated. On the fifth and sixth days, characterized as Stage 2, the muscle fatigue level induced by the two electrical currents will be evaluated. The first evaluation day will be divided into two phases. Phase 1 corresponds to the initial evaluation, anthropometric data collection and physical activity level evaluation. In Phase 2, the quadriceps femoris motor point will be located with a pen-shaped electrode and a neuromuscular electrical stimulation unit, and the subcutaneous adipose layer thickness covering the motor point will be evaluated by means of ultrasonography. Subsequently, the ultrasound probe will be maintained on the vastus lateralis muscle (VL) to obtain muscle architecture data at rest, during the maximal voluntary isometric contractions (MVICs) and during the evoked contractions. Next, a warming up protocol will be performed and the participants will perform three MVICs at the knee joint angles of 60° and 90° of knee flexion (0° = full knee extension) on the isokinetic dynamometer. Subsequently, the investigators will evaluate (1) the current intensity required to produce a torque equivalent to 20% MVIC, (2) the current intensity required to produce a 40 Nm torque, the maximum current intensity (mA) tolerated by the subject (3) at an angle of 60° of knee flexion, and (4) at 90° of knee flexion. From these evaluations, the investigators will analyze the neuromuscular efficiency (ratio between current intensity and evoked torque). After each NMES test, participants will indicate, on the visual-analog scale, the discomfort level perceived with each NMES current type. Clinical efficiency will be evaluated by the ratio between the discomfort level and the evoked torque in the above-described situations. On the second, third and fourth evaluation day, participants will perform all the evaluations described in Phase 2 of the first evaluation day, but with different configurations of the type of current randomized being applied. On the fifth day, the fatigue protocol will be applied with appropriated parameters according to the randomized current type, and sufficient current intensity to generate 20% of the MVIC. The discomfort level during the fatigue protocol will be recorded immediately after the end of the fatigue test. Participants will conduct three pre- and post-fatigue protocol MVICs in order to assess the fatigue level. For the sixth evaluation day, the same evaluations reported for the fifth day will be carried out, but with the second randomized current.

ELIGIBILITY:
Inclusion Criteria:

* Young male
* Age between 18 and 35 years
* Physically active,
* Normal knee function and range of motion
* No pain complaints
* No presence of lower limb pathology at the dominant limb.

Exclusion Criteria:

* Health problems (neurological, musculoskeletal impairment),
* Contraindication to maximal exercise,
* Having been treated with NMES in the last 3 months in the lower limb
* Not meeting the inclusion criteria.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary isometric contraction of the knee extensors | 14 minutes
  is an expression of the muscular strength, and will be evaluated by dynamometry.
Knee extensors evoked torque during the tests at submaximal current intensity levels | During 90 seconds of electrical stimulation
  is an expression describing the muscular strength generated by electrical stimulation, and will be assessed by dynamometry.
Knee extensors evoked torque during the tests at maximal current intensity levels | During 90 seconds of electrical stimulation
  is an expression describing the muscular strength generated by electrical stimulation, and will be assessed by dynamometry.
Knee extensors evoked torque during the fatigue protocol | During 20 minutes of electrical stimulation
  is an expression describing the muscular strength generated by electrical stimulation, and will be assessed by dynamometry.
Muscular architecture during the knee extensors maximum voluntary isometric contraction tests | 14 minutes
  is an expression used to describe the muscle fibers arrangement within the muscle, and is evaluated by determining the muscle thickness, fascicle pennation angle and fascicle length, which will be assessed by ultrasonography.
Muscular architecture during knee extensors evoked torque tests at submaximal current intensity levels | During 90 seconds of electrical stimulation
  is an expression used to describe the muscle fibers arrangement within the muscle, and is evaluated by determining the muscle thickness, fascicle pennation angle and fascicle length, which will be assessed by ultrasonography.
Muscular architecture during knee extensors evoked torque tests at maximal current intensity levels | During 90 seconds of electrical stimulation
  is an expression used to describe the muscle fibers arrangement within the muscle, and is evaluated by determining the muscle thickness, fascicle pennation angle and fascicle length, which will be assessed by ultrasonography.
Muscular architecture during the fatigue protocol | During 20 minutes of electrical stimulation
  is an expression used to describe the muscle fibers arrangement within the muscle, and is evaluated by determining the muscle thickness, fascicle pennation angle and fascicle length, which will be assessed by ultrasonography.
Discomfort level generated by electrical stimulation during evoked torque tests at submaximal current intensity levels | During 90 seconds of electrical stimulation
  Discomfort will be measured with a Visual Analogue Scale (0-100mm), where 0 and 100 mm corresponded to no discomfort and worst perceived discomfort, respectively.
Discomfort level generated by electrical stimulation during evoked torque tests at maximal current intensity levels | During 90 seconds of electrical stimulation
  Discomfort will be measured with a Visual Analogue Scale (0-100mm), where 0 and 100 mm corresponded to no discomfort and worst perceived discomfort, respectively.
Discomfort level generated by electrical stimulation during the fatigue protocol | During 20 minutes of electrical stimulation
  Discomfort will be measured with a Visual Analogue Scale (0-100mm), where 0 and 100 mm corresponded to no discomfort and worst perceived discomfort, respectively.
Current intensity required to evoke knee extensors submaximal torque | During 90 seconds of electrical stimulation
  Current intensity is defined as the amount or amplitude of electrical current (in milliamperes - mA) required to achieve a specific force, and will be evaluated in the electrical stimulation device.
Current intensity required to evoke knee extensors maximal torque | During 90 seconds of electrical stimulation
  Current intensity is defined as the amount or amplitude of electrical current (in milliamperes - mA) required to achieve a specific force, and will be evaluated in the electrical stimulation device.
Neuromuscular efficiency during knee extensors submaximal evoked torque tests | During 90 seconds of electrical stimulation
  Neuromuscular efficiency of the electrical currents will be evaluated by calculating the current intensity (input parameter or input) by the evoked torque (output parameter) ratio.
Neuromuscular efficiency during knee extensors maximal evoked torque tests | During 90 seconds of electrical stimulation
  Neuromuscular efficiency of the electrical currents will be evaluated by calculating the current intensity (input parameter or input) by the evoked torque (output parameter) ratio.
Neuromuscular efficiency during the fatigue protocol | During 20 minutes of electrical stimulation
  Neuromuscular efficiency of the electrical currents will be evaluated by calculating the current intensity (input parameter or input) by the evoked torque (output parameter) ratio.
Clinical efficiency during knee extensors submaximal evoked torque tests | During 90 seconds of electrical stimulation
  Clinical efficiency of the two electrical currents will be evaluated by calculating the ratio between the evoked torque (output parameter) and the level of discomfort generated.
Clinical efficiency during knee extensors maximal evoked torque tests | During 90 seconds of electrical stimulation
  Clinical efficiency of the two electrical currents will be evaluated by calculating the ratio between the evoked torque (output parameter) and the level of discomfort generated.
Clinical efficiency during the fatigue protocol | During 20 minutes of electrical stimulation
  Clinical efficiency of the two electrical currents will be evaluated by calculating the ratio between the evoked torque (output parameter) and the level of discomfort generated.
Muscle Fatigue Index | During 20 minutes of electrical stimulation
  Characterized by the force decrease after the fatigue protocol, it will be evaluated by dynamometry.
Fatigue Index from Evoked Torque | During 20 minutes of electrical stimulation
  Characterized by the decrease of the evoked torque during the fatigue protocol, the fatigue index from evoked torque will be evaluated by dynamometry, and obtained by the analysis of evoked torque curves.
Total work generated during the fatigue protocol | During 20 minutes of electrical stimulation
  The torque-time integral of the evoked torque curves during the fatigue protocol will be evaluated. The sum of the torque curve integral of all evoked contractions during the fatigue protocol will be calculated to determine the total work evoked by each current during the fatigue protocol.

SECONDARY OUTCOMES:
Thickness of the subcutaneous fat layer on the motor point | It will be evaluated during the first evaluation day.
  Corresponds to the amount of subcutaneous adipose tissue and will be evaluated by ultrasonography.
Level of physical activity | 8 minutes. It will be evaluated during the first evaluation day
  The level of physical activity (PA) of each subject will be assessed by the International Physical Activity Questionnaire (IPAQ).The scores will be assessed by calculating the metabolic equivalents (MET) for each activity level. Walking score will be achieved by the multiplication of 3.3 METs with the total walking duration in minutes in a week. Moderate physical activity scores will be achieved by the multiplication of 4.0 METs with the total moderate physical activity duration in minutes in a week. Vigorous physical activity scores will be achieved by the multiplication of 8.0 METs with the total vigorous physical activity duration in minutes in a week. Total physical activity MET-minutes/week will be obtained through sum of walking, moderate and vigorous MET minutes/week scores. Categorical Score will be classified into three levels of physical activity: low, moderate and high.

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paz IA, Rigo GT, Sgarioni A, Baroni BM, Frasson VB, Vaz MA. Alternating Current Is More Fatigable Than Pulsed Current in People Who Are Healthy: A Double-Blind, Randomized Crossover Trial. Phys Ther. 2021 Jun 1;101(6):pzab056. doi: 10.1093/ptj/pzab056. PMID 33561279